CLINICAL TRIAL: NCT04346485
Title: Prospective Randomized Comparison of SP TFL and Ho:YAG for RIRS Using 145 µm and 200 µm Fibers for the Management of Lower Pole Kidney Stones: Single-center Study
Brief Title: Comparison of SP TFL and Ho:YAG for RIRS Using 145 µm and 200 µm Fibers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy director for research, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sechenov-RIRS-20
Record Dates: First submitted 2020-03-12; First posted 2020-04-15 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Kidney Stone; Nephrolithiasis; Urolithiasis
Keywords: RIRS; holmium laser; superpulse thulium laser; kidney stone disease
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Urolithiasis | interventions — Dietary Fiber

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SP TFL RIRS with 145 mcm fiber (Experimental): Superpulse thulium fiber laser RIRS with 145 mcm laser fiber
  Interventions: Procedure: SP TFL RIRS with 145 mcm fiber
- SP TFL RIRS with 200 mcm fiber (Experimental): Superpulse thulium fiber laser RIRS with 200 mcm laser fiber
  Interventions: Procedure: SP TFL RIRS with 200 mcm fiber
- Ho:YAG RIRS with 200 mcm fiber (Active Comparator): Ho:YAG laser RIRS with 200 mcm laser fiber
  Interventions: Procedure: Ho:YAG RIRS with 200 mcm fiber

INTERVENTIONS:
Procedure: SP TFL RIRS with 145 mcm fiber — retrograde intrarenal surgery
  Arms: SP TFL RIRS with 145 mcm fiber
Procedure: SP TFL RIRS with 200 mcm fiber — retrograde intrarenal surgery
  Arms: SP TFL RIRS with 200 mcm fiber
Procedure: Ho:YAG RIRS with 200 mcm fiber — retrograde intrarenal surgery
  Arms: Ho:YAG RIRS with 200 mcm fiber

SUMMARY:
The authors hypothesize that the RIRS using 150-microm Tm-fiber laser is superior than fiber with larger diameters, as 200-microm Tm-fiber laser or 200-microm holmium fiber laser, in such points as follows:

* decreasing surgery time and laser-on time due to possibility of 4.3 fold ablation efficacy increase, which has been shown by Andreeva et al.;
* increasing the flexible ureteroscope tip deflection lower pole stones availability;
* decreased risk of complications and a better irrigation and visualization due to better irrigation with smaller fiber;
* increasing of lithotripsy efficacy and laser beam density by lowering of beam focal spot due to using of lesser fiber diameter

DETAILED DESCRIPTION:
RIRS will be performed with SP TFL or Ho:YAG (100 W). The procedure is performed under general anesthesia with the patient in the dorsal lithotomy position. The bladder is entered either with a cystoscope or a semi-rigid ureterorenoscope. Guidewires (0.035") will be used to facilitate access (under fluoroscopic guidance). After access sheath (12/14) will be placed up to the kidney pelvis. Through the access sheath ureteroscope will be introduced. For nephrolithotripsy 145 mcm and 200 mcm fibers will be used. Large fragments could be extracted with nitinol basket. After the surgery ureteral stent (7 Fr.) will be placed inside the ureter for 10 to 14 days.

A 10 Fr urethral catheter can be placed in the bladder for the drainage of the bladder during the operation.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females > 18 y.o.;
* Radiologically confirmed (CT) kidney stone;
* Stone size from 10 to 20 mm.

Exclusion Criteria:

• Multiple (more than 3) kidney stones > 5 mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Laser-on time | during surgery
  Time of laser emission during surgery, seconds

SECONDARY OUTCOMES:
adverse events | during surgery and 6 months after surgery
  Complications according to Clavien-Dindo classification (higher score means more severe complication)
Operative time | during surgery
  Surgery duration, minutes
Hemoglobin drop | 1 day after surgery
  Change of hemoglobin level 1 day after surgery comparing to pre-operative value, g/L
Catheter stay | 1 week
  duration of catheterisation, days
hospitalization length | 1 week
  Duration of hospital stay after surgery, days
Radiation exposure | during surgery
  Duration of X-ray exposure, sec.
Radiation exposure | during surgery
  Effective dose, mSv
Stone-free rate | 3 month
  Percentage of patients with absence of stones larger 3 mm in maximum size on follow-up CT

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Urology and Reproductive Health, Sechenov University., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No